CLINICAL TRIAL: NCT01496235
Title: Randomized Clinical Trial of the Effect of Cocoa Consumption in Cardiovascular and Immune Parameters in Colombian Patients With Newly Diagnosed Stage 1 Arterial Hypertension
Brief Title: Effect of Cocoa Consumption in Cardiovascular and Immune Parameters
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties with the patient recruitment
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Monica Lucia Giraldo, Principal Investigator, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Cacao I
Record Dates: First submitted 2011-11-24; First posted 2011-12-21 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Arterial Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dark chocolate (Active Comparator): Presence of 70% cocoa solids
  Interventions: Dietary Supplement: Dark chocolate
- White chocolate (Placebo Comparator)
  Interventions: Dietary Supplement: White chocolate

INTERVENTIONS:
Dietary Supplement: Dark chocolate — Each chocolate bar provided 210 calories represented in 25 grams of carbohydrates, 3 g of proteins, 18 g of total fat and the presence of 70% cocoa solids
  Arms: Dark chocolate
Dietary Supplement: White chocolate — Each chocolate bar provided 230 calories represented in 28 grams of carbohydrates, 3 g of proteins, 18 g of total fat, without the presence of 70% cocoa solids
  Arms: White chocolate

SUMMARY:
Arterial hypertension is one of the most preventable risk factors for stroke, cardiovascular and renal disease. Cocoa is rich in a subclass of flavonoid called flavanol this increase nitric oxide production and is involved in controlling blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 65 years old
* Resides in Medellín City
* Attached from the contributive regimen of Colombian Health System
* Essential Arterial Hypertension, stage I. Diagnosis less than 3 months.
* Medically indicated non-pharmacological therapy.
* Voluntary desire to consume 50 grams of chocolate per day for 12 weeks.
* Voluntary desire to participate in the trial and sign informed consent.

Exclusion Criteria:

* Suspect of secondary hypertension
* Suspect of injury in target organ
* Presence of diabetes mellitus
* BMI (Body Mass Index) major or equal to 30
* Present smoker or with less than four weeks of abstinence of tobacco
* Consume antiplatelet substances
* Regular consumption of antioxidants, multivitamins, anti-inflammatory medications, drugs for nasal congestion and sibutramine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2009-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in diastolic blood pressure | Baseline and 12 weeks
  Measurement of the diastolic blood pressure with the ambulatory blood pressure monitoring

SECONDARY OUTCOMES:
Change in systolic blood pressure | Baseline and 12 weeks
  Measurement of the systolic blood pressure with the ambulatory blood pressure monitoring
Change in total cholesterol | Baseline and 12 weeks
Change in low density lipoprotein cholesterol | Baseline and 12 weeks
Change in high density lipoprotein cholesterol | Baseline and 12 weeks
Change in triglycerides levels | Baseline and 12 weeks
Change in hs-CRP | Baseline and 12 weeks
Change in IL-1 beta levels | Baseline and 12 weeks
Change in IL-2 levels | Baseline and 12 weeks
Change in tumor necrosis factor alpha levels | Baseline and 12 weeks
Change in flow mediated dilatation of the brachial artery | Baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Monica L Giraldo, PhD, Principal Investigator — Universidad de Antioquia
Locations (1):
- Sede Investigaciones Universitarias, Universidad de Antioquia, Medellín, Antioquia, Colombia

REFERENCES:
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. National Heart, Lung, and Blood Institute; National High Blood Pressure Education Program Coordinating Committee. Seventh report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. Hypertension. 2003 Dec;42(6):1206-52. doi: 10.1161/01.HYP.0000107251.49515.c2. Epub 2003 Dec 1. PMID 14656957
- [Background] Mancia G, De Backer G, Dominiczak A, Cifkova R, Fagard R, Germano G, Grassi G, Heagerty AM, Kjeldsen SE, Laurent S, Narkiewicz K, Ruilope L, Rynkiewicz A, Schmieder RE, Boudier HA, Zanchetti A; ESH-ESC Task Force on the Management of Arterial Hypertension. 2007 ESH-ESC Practice Guidelines for the Management of Arterial Hypertension: ESH-ESC Task Force on the Management of Arterial Hypertension. J Hypertens. 2007 Sep;25(9):1751-62. doi: 10.1097/HJH.0b013e3282f0580f. No abstract available. PMID 17762635
- [Background] K Hollenberg N. Vascular action of cocoa flavanols in humans: the roots of the story. J Cardiovasc Pharmacol. 2006;47 Suppl 2:S99-102; discussion S119-21. doi: 10.1097/00005344-200606001-00002. PMID 16794463
- [Background] McCullough ML, Chevaux K, Jackson L, Preston M, Martinez G, Schmitz HH, Coletti C, Campos H, Hollenberg NK. Hypertension, the Kuna, and the epidemiology of flavanols. J Cardiovasc Pharmacol. 2006;47 Suppl 2:S103-9; discussion 119-21. doi: 10.1097/00005344-200606001-00003. PMID 16794446
- [Background] Keen CL, Holt RR, Oteiza PI, Fraga CG, Schmitz HH. Cocoa antioxidants and cardiovascular health. Am J Clin Nutr. 2005 Jan;81(1 Suppl):298S-303S. doi: 10.1093/ajcn/81.1.298S. PMID 15640494
- [Background] Selmi C, Mao TK, Keen CL, Schmitz HH, Eric Gershwin M. The anti-inflammatory properties of cocoa flavanols. J Cardiovasc Pharmacol. 2006;47 Suppl 2:S163-71; discussion S172-6. doi: 10.1097/00005344-200606001-00010. PMID 16794453
- [Background] Desch S, Schmidt J, Kobler D, Sonnabend M, Eitel I, Sareban M, Rahimi K, Schuler G, Thiele H. Effect of cocoa products on blood pressure: systematic review and meta-analysis. Am J Hypertens. 2010 Jan;23(1):97-103. doi: 10.1038/ajh.2009.213. Epub 2009 Nov 12. PMID 19910929
- [Background] Ried K, Sullivan T, Fakler P, Frank OR, Stocks NP. Does chocolate reduce blood pressure? A meta-analysis. BMC Med. 2010 Jun 28;8:39. doi: 10.1186/1741-7015-8-39. PMID 20584271
- [Background] Taubert D, Roesen R, Schomig E. Effect of cocoa and tea intake on blood pressure: a meta-analysis. Arch Intern Med. 2007 Apr 9;167(7):626-34. doi: 10.1001/archinte.167.7.626. PMID 17420419
- [Background] Grassi D, Necozione S, Lippi C, Croce G, Valeri L, Pasqualetti P, Desideri G, Blumberg JB, Ferri C. Cocoa reduces blood pressure and insulin resistance and improves endothelium-dependent vasodilation in hypertensives. Hypertension. 2005 Aug;46(2):398-405. doi: 10.1161/01.HYP.0000174990.46027.70. Epub 2005 Jul 18. PMID 16027246
- [Background] Sabater-Hernandez D, Fikri-Benbrahim O, Faus MJ. [Usefulness of ambulatory blood pressure monitoring for clinical decisions making]. Med Clin (Barc). 2010 Jun 5;135(1):23-9. doi: 10.1016/j.medcli.2009.07.019. Epub 2009 Oct 12. Spanish. PMID 19819484
- [Background] Haukoos JS, Newgard CD. Advanced statistics: missing data in clinical research--part 1: an introduction and conceptual framework. Acad Emerg Med. 2007 Jul;14(7):662-8. doi: 10.1197/j.aem.2006.11.037. Epub 2007 May 30. PMID 17538078
- [Background] Farouque HM, Leung M, Hope SA, Baldi M, Schechter C, Cameron JD, Meredith IT. Acute and chronic effects of flavanol-rich cocoa on vascular function in subjects with coronary artery disease: a randomized double-blind placebo-controlled study. Clin Sci (Lond). 2006 Jul;111(1):71-80. doi: 10.1042/CS20060048. PMID 16551272
- [Background] Crews WD Jr, Harrison DW, Wright JW. A double-blind, placebo-controlled, randomized trial of the effects of dark chocolate and cocoa on variables associated with neuropsychological functioning and cardiovascular health: clinical findings from a sample of healthy, cognitively intact older adults. Am J Clin Nutr. 2008 Apr;87(4):872-80. doi: 10.1093/ajcn/87.4.872. PMID 18400709
- [Background] Monagas M, Khan N, Andres-Lacueva C, Casas R, Urpi-Sarda M, Llorach R, Lamuela-Raventos RM, Estruch R. Effect of cocoa powder on the modulation of inflammatory biomarkers in patients at high risk of cardiovascular disease. Am J Clin Nutr. 2009 Nov;90(5):1144-50. doi: 10.3945/ajcn.2009.27716. Epub 2009 Sep 23. PMID 19776136
- [Background] Engler MB, Engler MM, Chen CY, Malloy MJ, Browne A, Chiu EY, Kwak HK, Milbury P, Paul SM, Blumberg J, Mietus-Snyder ML. Flavonoid-rich dark chocolate improves endothelial function and increases plasma epicatechin concentrations in healthy adults. J Am Coll Nutr. 2004 Jun;23(3):197-204. doi: 10.1080/07315724.2004.10719361. PMID 15190043
- [Background] Muniyappa R, Hall G, Kolodziej TL, Karne RJ, Crandon SK, Quon MJ. Cocoa consumption for 2 wk enhances insulin-mediated vasodilatation without improving blood pressure or insulin resistance in essential hypertension. Am J Clin Nutr. 2008 Dec;88(6):1685-96. doi: 10.3945/ajcn.2008.26457. PMID 19064532
- [Background] Taubert D, Roesen R, Lehmann C, Jung N, Schomig E. Effects of low habitual cocoa intake on blood pressure and bioactive nitric oxide: a randomized controlled trial. JAMA. 2007 Jul 4;298(1):49-60. doi: 10.1001/jama.298.1.49. PMID 17609490
- [Background] Grassi D, Desideri G, Necozione S, Lippi C, Casale R, Properzi G, Blumberg JB, Ferri C. Blood pressure is reduced and insulin sensitivity increased in glucose-intolerant, hypertensive subjects after 15 days of consuming high-polyphenol dark chocolate. J Nutr. 2008 Sep;138(9):1671-6. doi: 10.1093/jn/138.9.1671. PMID 18716168
- [Background] Fraga CG, Actis-Goretta L, Ottaviani JI, Carrasquedo F, Lotito SB, Lazarus S, Schmitz HH, Keen CL. Regular consumption of a flavanol-rich chocolate can improve oxidant stress in young soccer players. Clin Dev Immunol. 2005 Mar;12(1):11-7. doi: 10.1080/10446670410001722159. PMID 15712594
- [Background] Wang-Polagruto JF, Villablanca AC, Polagruto JA, Lee L, Holt RR, Schrader HR, Ensunsa JL, Steinberg FM, Schmitz HH, Keen CL. Chronic consumption of flavanol-rich cocoa improves endothelial function and decreases vascular cell adhesion molecule in hypercholesterolemic postmenopausal women. J Cardiovasc Pharmacol. 2006;47 Suppl 2:S177-86; discussion S206-9. doi: 10.1097/00005344-200606001-00013. PMID 16794456
- [Background] Holt RR, Actis-Goretta L, Momma TY, Keen CL. Dietary flavanols and platelet reactivity. J Cardiovasc Pharmacol. 2006;47 Suppl 2:S187-96; discussion S206-9. doi: 10.1097/00005344-200606001-00014. PMID 16794457
- [Background] Murphy KJ, Chronopoulos AK, Singh I, Francis MA, Moriarty H, Pike MJ, Turner AH, Mann NJ, Sinclair AJ. Dietary flavanols and procyanidin oligomers from cocoa (Theobroma cacao) inhibit platelet function. Am J Clin Nutr. 2003 Jun;77(6):1466-73. doi: 10.1093/ajcn/77.6.1466. PMID 12791625
- [Background] Ferri C, Grassi D, Grassi G. Cocoa beans, endothelial function and aging: an unexpected friendship? J Hypertens. 2006 Aug;24(8):1471-4. doi: 10.1097/01.hjh.0000239279.82196.ec. No abstract available. PMID 16877946
- [Background] Schroeter H, Heiss C, Balzer J, Kleinbongard P, Keen CL, Hollenberg NK, Sies H, Kwik-Uribe C, Schmitz HH, Kelm M. (-)-Epicatechin mediates beneficial effects of flavanol-rich cocoa on vascular function in humans. Proc Natl Acad Sci U S A. 2006 Jan 24;103(4):1024-9. doi: 10.1073/pnas.0510168103. Epub 2006 Jan 17. PMID 16418281
- [Background] Hermann F, Spieker LE, Ruschitzka F, Sudano I, Hermann M, Binggeli C, Luscher TF, Riesen W, Noll G, Corti R. Dark chocolate improves endothelial and platelet function. Heart. 2006 Jan;92(1):119-20. doi: 10.1136/hrt.2005.063362. No abstract available. PMID 16365364